CLINICAL TRIAL: NCT05599997
Title: Investigation of Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of a Single Oral Dose of 30 mg BAY 1753011 Given as IR Tablet in Male and Female Participants in a Multicenter, Non-randomized, Non-controlled, Non-blinded Study With Group Stratification in Participants With Renal Impairment and Control Group Matched for Age-, Gender-, and Weight
Brief Title: A Study to Learn How the Study Treatment BAY1753011 Moves Into, Through and Out of the Body, How it Works, How Safe it is, and How it Affects the Body When Given Once as Tablet in Male and Female Participants With Reduced Kidney Function Compared to Matched Participants With Normal Kidney Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 19482; 2019-000876-41 (EudraCT Number)
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Congestive Heart Failure; Renal Impairment
MeSH Terms: conditions — Heart Failure; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy (Experimental): Age-, weight- and gender- matched control group of healthy volunteers received a single oral dose of 30 mg BAY1753011 tablet.
  Interventions: Drug: Pecavaptan (BAY1753011)
- Mild renal impairment (Experimental): Subjects with mild renal impairment received a single oral dose of 30 mg BAY1753011 tablet.
  Interventions: Drug: Pecavaptan (BAY1753011)
- Moderate renal impairment (Experimental): Subjects with moderate renal impairment received a single oral dose of 30 mg BAY1753011 tablet.
  Interventions: Drug: Pecavaptan (BAY1753011)
- Severe renal impairment (Experimental): Subjects with severe renal impairment received a single oral dose of 15 mg BAY1753011 tablet.
  Interventions: Drug: Pecavaptan (BAY1753011)

INTERVENTIONS:
Drug: Pecavaptan (BAY1753011) — 30 mg, immediate release tablet, single dose, oral
  Arms: Healthy; Mild renal impairment; Moderate renal impairment
Drug: Pecavaptan (BAY1753011) — 15 mg, immediate release tablet, single dose, oral
  Arms: Severe renal impairment

SUMMARY:
Researchers are looking for a better way to treat people with heart failure. Heart failure is a condition which occurs when the heart does not pump blood as well as it should leading to shortness of breath, tiredness, and ankle swelling.

The study treatment BAY1753011 is under development to treat heart failure. It is thought to reduce the action of a hormone called vasopressin that is naturally produced in the body. People with heart failure often have elevated levels of vasopressin. This is known to result in worsening of the heart failure condition.

People with heart failure often also have reduced kidney functions. As kidneys play a role in removal of drugs from the body, reduced kidney function may result in higher blood levels of BAY1753011.

The main purpose of this study was to learn how BAY1753011 moved into, through and out of the body in participants with different degrees of reduced kidney function compared to matched participants (age, gender, and weight) with normal kidney function.

To answer this, the researchers compared:

* the (average) total level of BAY1753011 in the blood (also called AUC)
* the (average) highest level of BAY1753011 in the blood (also called Cmax) between the different groups with reduced kidney function (mild/moderate/severe) and the control group (normal kidney function).

In addition, the researchers wanted to know how safe BAY1753011 was and the degree to which overt medical problems caused by it could be tolerated (also called tolerability) by the different groups of participants.

These medical problems are also known as "adverse events". Doctors keep track of all medical problems that happen in studies, even if they do not think they might be related to the study treatments.

All participants took a single dose of BAY1753011 in tablet form by mouth. Each participant was in the study for approximately 3 to 4 weeks, including an in-house phase of 5 days and 4 nights with one treatment day.

During the study, the doctors and their study team:

* did physical examinations
* checked vital signs such as blood pressure, heart rate, body temperature and number of breaths within a minute (respiratory rate)
* examined heart health using electrocardiogram (ECG)
* took blood and urine samples
* counted the number of toilet visits during the night

ELIGIBILITY:
Inclusion Criteria:

* Male or female White participants (women without childbearing potential)
* Aged from ≥18 years
* body mass index above or equal 18.5 kg/m2 and below or equal 36 kg/m2 at the first screening visit
* Participants with renal impairment: with an eGFR <90 mL/min/1.73 m^2 determined from serum creatinine 21-3 days prior to dosing using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
* Age-, weight- and gender- matched control group

Exclusion Criteria:

* An anatomical abnormality of the gut that could affect the retention times of the drug in the stomach/gut adversely
* Conditions or concomitant treatment that might adversely affect the gastric pH level
* Pancreatic dysfunction/insufficiency
* Febrile illness within 4 week prior to admission to study center
* Known hypersensitivity to the study drugs
* Known severe allergies, non-allergic drug reactions, or multiple drug allergies
* Participants with a medical disorder, condition or history of such that would impair the participant's ability to participate or complete this study in the opinion of the investigator or the Sponsor
* Concomitant treatment from 2 weeks before study drug administration until end of follow-up with drugs that may impact the PK of BAY 1753011:Strong and moderate inducers or inhibitors of CYP3A4Moderate and strong inhibitors of P-gp transport Probenecid and valproic acid
* Concomitant treatment with potassium-sparing diuretic (with the exception of mineralocorticoid- receptor antagonist [MRA]) that cannot be stopped prior to randomization and for the duration of the treatment period
* Although no clinical study data are available for BAY 1753011, drugs for the treatment of hyperphosphatemia such as sevelamer or lanthanum should not be given from 24 h before until 24 h after dosing, as they are known to bind many anionic drugs
* Acute renal failure
* Active nephritis
* Severe infection or any clinically significant illness within 4 weeks prior to dosing
* Impairment of any other major organ system other than the kidney
* Clinically relevant findings in the ECG such as a second- or third-degree atrioventricular (AV) block, prolongation of the QTc-interval over 480 msec
* Systolic blood pressure below 100 or above 160 mmHg
* Diastolic blood pressure below 50 or above 100 mmHg
* Heart rate below 50 or above 100 beats/ min

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2021-01-22 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Area under the concentration versus time curve from zero to infinity divided by dose of total BAY1753011 in plasma after single dose administration (AUC/D) | From pre-dose until 144 hours post dose
  Dose-normalized AUC (AUC/D) of BAY1753011 was investigated as the dose for the severe renal impairment group was reduced to 15 mg.
Maximum observed drug concentration divided by dose of total BAY1753011 in plasma after single dose administration (Cmax/D) | From pre-dose until 144 hours post dose
  Dose-normalized Cmax (Cmax/D) of BAY1753011 was investigated as the dose for the severe renal impairment group was reduced to 15 mg.
Area under the concentration versus time curve from zero to infinity divided by dose of unbound BAY1753011 in plasma after single dose administration (AUCu/D) | From pre-dose until 144 hours post dose
  Dose-normalized AUCu (AUCu/D) of BAY1753011 was investigated as the dose for the severe renal impairment group was reduced to 15 mg.
Maximum observed drug concentration divided by dose of unbound BAY1753011 in plasma after single dose administration (Cmax,u/D) | From pre-dose until 144 hours post dose
  Dose-normalized Cmax,u (Cmax,u/D) of BAY1753011 was investigated as the dose for the severe renal impairment group was reduced to 15 mg.

SECONDARY OUTCOMES:
Number of participants with treatment-emergent adverse events | After first application of study medication up to 10 days after the study medication

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - APEX GmbH, München, Bavaria
  - CRS Clinical-Research-Services Kiel GmbH, Kiel, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.